CLINICAL TRIAL: NCT02620124
Title: GnRH Anonist as Luteal Support in Frozen-thawed Embryo Transfer Cycles
Brief Title: GnRH Agonist as Luteal Support in FET Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T5/2013
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Natural cycle, control (No Intervention): Treatment cycles with normal luteal support with progesteron
- Natural cycle, intervention (Experimental): Treatment cycles with normal luteal support with progesteron and a single dose of 0.1 mg triptorelin when the age of the embryo was 6 days: Intervention is the additional 0.1 mg triptorelin as described in the previous sentence.
  Interventions: Drug: Natural cycle: Triptorelin acetate 0.1 mg
- Hormone replacement cycle, control (No Intervention): Standard hormone replacement cycle with estrogen and progesteron
- Hormone replacement cycle, intervention (Experimental): Standard hormone replacement cycle with estrogen and progesteron and a single dose of 0.1 mg triptorelin when the age of the embryo was 6 days
  Interventions: Drug: Natural cycle: Triptorelin acetate 0.1 mg; Drug: Hormone replacement cycle and triptorelin acetate 0.1 mg

INTERVENTIONS:
Drug: Natural cycle: Triptorelin acetate 0.1 mg — A single dose of triptorelin acetate 0.1 s.c. was giwen when the age of the transferred embryo was six days in additon to standard micronized progesterone 400 mg vaginally
  Arms: Hormone replacement cycle, intervention; Natural cycle, intervention
Drug: Hormone replacement cycle and triptorelin acetate 0.1 mg — A single dose of triptorelin acetate 0.1 s.c. was giwen when the age of the transferred embryo was six days in addition to standard Estradiol and progesterone support
  Arms: Hormone replacement cycle, intervention

SUMMARY:
Back ground: A single dose of GnRH analogue in the luteal phase is reported to improve the outcome of IVF/ICSI treatments but the effect in FET cycles has not been reported.

Aim: To compare the results of frozen thawed embryo transfers with and without GnRHa analogue support Primary end point: IR, PR, on going PR Secondary end point: hCH, E2 and progesterone levels 14 days after thawing

ELIGIBILITY:
Inclusion Criteria:

* 20 - 45 year old women comig to frozen thawed embryo transfer

Exclusion Criteria:

* The age of the woman over 42 years during the initial ICF/ICSI- treatment from which the embryos derive
* Abnormal uterus
* Known abnormality of karyotype of the woman or her partner
* Severe male factor as an exclusive reason for subfertility
* Allegy for triptorelin acetate

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | five weeks after the embryo transfer
Implantation rate | five weeks after the embryo transfer
Ongoing pregnancy rate | ten weeks after the embryo transfer

SECONDARY OUTCOMES:
hCG- level | 14 days after thawing of the embryos

CONTACTS AND LOCATIONS:
Overall Officials: Varpu Jokimaa, MD, PhD, Principal Investigator — Hospital District of the South-West Finland

IPD SHARING:
Plan to Share IPD: No